CLINICAL TRIAL: NCT04837807
Title: Understanding Quality of Life in High Digital Device Users Who Are Treated With Systane Hydration PF
Brief Title: Digital Device Users Who Are Treated With Systane Hydration PF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Andrew Pucker, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-30007063
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Results first posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Dry Eye
Keywords: Digital Eye Strain; Dry Eye; Artificial Tears; Eye Comfort
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: All subjects will be treated with Systane Hydration PF. Half will start with the unit-dose version and half with start with the multi-dose version. Subjects will switch to the other dosing option in the middle of the study.
Who Masked: Participant
Masking Description: Investigators will be masked to the dosage group. Subjects will not be masked because it is not possible with the dosage interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Unit Dose First, Then Multi-Dose (Experimental): Subjects randomized to this group will apply the unit-dose version of Systane Hydration PF to determine if it helps alleviate symptoms associated with digital eye strain.
  Interventions: Drug: Systane Hydration PF
- Multi Dose, Then Unit Dose (Experimental): Subjects randomized to this group will apply multi-dose version of Systane Hydration PF to determine if it helps alleviate symptoms associated with digital eye strain.
  Interventions: Drug: Systane Hydration PF

INTERVENTIONS:
Drug: Systane Hydration PF — This is an over-the-counter preservative free artificial tear that can be purchased at most retail stores and pharmacies.

SUMMARY:
Systane Hydration PF is a recently released preservative-free artificial tear that is able to supplement the ocular surface's moisture while simultaneously soothing the eye. While Systane Hydration PF should in theory improve the symptoms and subsequently the quality of life of patients who have DES, this clinical application has yet to be tested. This drop furthermore is available in both unit-dose and multi-dose options; however, it is unclear if patient perceive a difference between the two dispensing methods. Therefore, the primary purpose of this study is to recruit patients who have DES and to treat them with Systane Hydration PF and determine how regular use of this drop impacts a patient's ocular surface symptoms and overall quality of life. This study will secondarily compare the two dispensing methods to determine if patients prefer one method over the other.

DETAILED DESCRIPTION:
Extensive computer use is no longer an employment-specific challenge. Use of digital devices in work, home, and leisure settings is now the norm, and it is now socially expected. While the introduction of high-powered computers and digital devices have greatly improved many aspects of modern life, the pervasive use of digital devices has caused some patients to develop a condition known as Digital Eye Strain (DES). DES has been reported to be as high as 93% the population depending upon how the condition is defined, and its severity has been found to increase with increased digital device time. DES is a condition where patients experience symptoms such as glare, accommodative dysfunction, defocus, fatigue, discomfort, and dryness from digital device use, and these dry eye symptoms may also result in decreased quality of life. While dryness symptoms in DES are likely multifactorial (e.g., contact lens use, systemic disease status), much of the dryness symptoms in DES are probably due to tear film evaporation secondary to having a reduced number of blinks per minute while using digital devices. Since much of the ocular symptoms associated with DES stem from excessive tear evaporation, artificial tears have become an accepted DES treatment

Systane Hydration PF is a recently released preservative-free artificial tear that is able to supplement the ocular surface's moisture while simultaneously soothing the eye. Systane Hydration PF has HydroBoost technology, which is thought to enhance the drop's effectiveness by incorporating ingredients that increase drop retention. While Systane Hydration PF should in theory improve the symptoms and subsequently the quality of life of patients who have DES, this clinical application has yet to be tested. This drop furthermore is available in both unit-dose and multi-dose options; however, it is unclear if patient perceive a difference between the two dispensing methods. Therefore, the primary purpose of this study is to recruit patients who have DES and to treat them with Systane Hydration PF and determine how regular use of this drop impacts a patient's ocular surface symptoms and overall quality of life. This study will secondarily compare the two dispensing methods to determine if patients prefer one method over the other.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Using digital devices 8 or more hours per day
* Eyes that are dry, irritated, itchy or burn while using a digital screen, like a computer or smartphone
* Eye fatigue from digital screen use
* Impact of Dry Eye on Daily Life (IDEEL) Work score ≤80
* Ocular Surface Disease Index (OSDI) score between 13 and 32 (inclusive)
* Willing to discontinue current artificial tears for at least 24 hours before enrollment

Exclusion Criteria:

* Pregnant or breastfeeding
* Are currently using isotretinoin-derivatives or other ocular medications
* Having any active ocular infection or inflammation
* History of severe ocular trauma
* Ocular surgery within the past 12 months
* Having any known systemic health conditions that are thought to alter tear film physiology (e.g., Sjögren's syndrome
* Using a dry eye treatment other than artificial tears
* Currently using artificial tears more than 4 times per day
* Contact lens wear within the past week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Unit Dose, Then Multi-dose: The participants first received the unit dose version of Systane Hydrataion PF, there was a one day washout period, and then they received the multi-dose version of Systane Hydration PF.
- Multi Dose, Then Unit Dose: The participants first received the multi-dose version of Systane Hydrataion PF, there was a one day washout period, and then they received the unit-dose version of Systane Hydration PF.
Period: First Sequence (Week 1)
Arm/Group | Unit Dose, Then Multi-dose | Multi Dose, Then Unit Dose
Started (This was a crossover study, so all subject got both treatments.) | 15 | 15
Received Sequence | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout 1 Day
Arm/Group | Unit Dose, Then Multi-dose | Multi Dose, Then Unit Dose
Started | 15 | 14
Completed | 14 | 14
Not Completed | 1 | 0
Period: Second Sequence (Week 2)
Arm/Group | Unit Dose, Then Multi-dose | Multi Dose, Then Unit Dose
Started | 14 | 14
Completed (Person dropped out prior to the crossover.) | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Subjects were randomized to either a multi dose group or a unit dose group, each group used either a multi dose or unit does in order to apply Systane Hydration PF to determine if it helps alleviate symptoms associated with digital eye strain. After 1 week subjects were switched from their starting group to the other group to determine which dispensing method was preferred.
  Systane Hydration PF: This is an over-the-counter preservative free artificial tear that can be purchased at most retail stores and pharmacies.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: Years] | 28.6 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This project featured a total of 30 participants, each participant received both treatments, however one patient was lost to follow up, and thus was not part of the crossover total.
  Participants
    Female | 21
    Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: The project features only 30 participants, all participants got both treatments however one subject dropped out prior to the crossover and thus was not counted in the crossover total.
  participants
    United States | 30

OUTCOME MEASURES:

1. Primary Outcome: IDEEL (Impact of Dry Eye on Daily Life) Quality of Life - Work Subsection
Description: Impact of Dry Eye on Daily Life (IDEEL) Work questions will be self-administered electronically to understand how treatment with Systane Hydration PF helps a patient's ability to work (0-100 scale with 100 being worst and 0 being best).
Time Frame: 2 weeks
Population: While we had 30 total subjects enroll we lost one person due to lack of interest in the study. As such she was not switched over to the next group and thus no scores other than baseline were collected.
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- Unit Dose: Subjects randomized to this group will apply the unit-dose version of Systane Hydration PF to determine if it helps alleviate symptoms associated with digital eye strain.
  Systane Hydration PF: This is an over-the-counter preservative free artificial tear that can be purchased at most retail stores and pharmacies.
- Multi Dose: Subjects randomized to this group will apply multi-dose version of Systane Hydration PF to determine if it helps alleviate symptoms associated with digital eye strain.
  Systane Hydration PF: This is an over-the-counter preservative free artificial tear that can be purchased at most retail stores and pharmacies.
Arm/Group | Unit Dose | Multi Dose
Number analyzed (Participants) | 30 | 30
score on a scale | 81.4 (12.7) | 81.4 (12.7)
Statistical Analysis 1: Comparison: Unit Dose vs Multi Dose; Each participant in the study was asked to complete the IDEEL work at their baseline, week 1 and week 2 visits. The IDEEL work is graded on a scale to 100 with higher numbers being deemed as "better" scores thus representing more comfort than previous weeks; Test type: Superiority; p < 0.05, ANOVA; This was a cross-over study, so there is really 30 subjects per group that was analyzed; Mean Difference (Final Values) = 22.4, Standard Deviation 12.8

2. Secondary Outcome: Drop Dispensing Method Preference
Description: Subjects will report whether they preferred the unit-dose dispensing method or the multi-dose dispensing method via a forced choice questionnaire (forced choice with patient being required to pick if they like the unit-dose dispensing method or the multi-dose better).
Time Frame: Between groups at 2 weeks
Population: One person discontinued after the baseline visit and thus did not crossover between groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Unit Dose | Multi Dose
Number analyzed (Participants) | 29 | 29
Participants | 16 | 13

3. Secondary Outcome: Ocular Surface Disease Index (OSDI) Questionnaire
Description: The Ocular Surface Disease Index (OSDI) will be self-administered electronically to understand how treatment with Systane Hydration PF helps a patient's ability to work (0-100 scale with 100 being worst and 0 being best).
Time Frame: 2 weeks
Population: One subject was lost after the baseline visit. Thus OSDI scores for the week 1 and 2 visit could not be calculated for that individual.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unit Dose | Multi Dose
Number analyzed (Participants) | 29 | 30
score on a scale | 14.3 (8.6) | 14.3 (8.6)
Statistical Analysis 1: Comparison: Unit Dose vs Multi Dose; Test type: Superiority — OSDI scores were obtained across all three visits, baseline, week 1 and week 2. Lower OSDI scores indicate better eye health; p < 0.05, ANOVA; This was a cross-over study, so there is really 30 subjects per group that was analyzed; Mean Difference (Final Values) = 10.5, Standard Deviation 7.3

ADVERSE EVENTS:
Time Frame: 1 month.
Arm/Group | Unit Dose | Multi Dose
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT04837807/Prot_SAP_ICF_000.pdf